CLINICAL TRIAL: NCT02508688
Title: Thoracoscopic Mesh Repair of Diaphragmatic Defects for Hepatic Hydrothorax: 10 Years' Experience From a Single Large-volume Center
Brief Title: Thoracoscopic Mesh Repair of Diaphragmatic Defects for Hepatic Hydrothorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201506012RIND
Record Dates: First submitted 2015-07-21; First posted 2015-07-27 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Liver Cirrhosis
Keywords: hepatic hydrothorax; thoracoscopic surgery; diaphragmatic defect
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- thoracoscopic mesh repair group (Experimental): 63 patients with refractory HH (> 3 times thoracentesis and failure to maximal doses of diuretics) who underwent thoracoscopic diaphragmatic repair were included in this study.
  Interventions: Procedure: thoracoscopic diaphragmatic repair

INTERVENTIONS:
Procedure: thoracoscopic diaphragmatic repair — patients with refractory hepatic hydrothorax (> 3 times thoracentesis and failure to maximal doses of diuretics) who underwent thoracoscopic diaphragmatic repair

SUMMARY:
The management of refractory hepatic hydrothorax is challenging and usually unsuccessful. The study will discuss the perioperative treatment, effectiveness, and morphology of diaphragmatic defects of hepatic hydrothorax in thoracoscopic mesh repair. Risk factors associated with increased three-month mortality in these critically ill patients will be studied.

DETAILED DESCRIPTION:
Objective The objective was to analyze the outcomes of thoracoscopic mesh repair for hepatic hydrothorax (HH) at the institution of the investigators during the past 10 years.

Methods A total of 63 patients with refractory HH, who underwent thoracoscopic mesh onlay reinforcement to repair diaphragmatic defects from January 2005 to December 2014, were included in the study. Mesh covering alone was used in 47 patients and mesh with suturing was used in 16 patients. Patient demographics, Child-Pugh class, and model for end-stage liver disease (MELD) score were evaluated to predict morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* patients with refractory hepatic hydrothorax (> 3 times thoracentesis and failure to maximal doses of diuretics)

Exclusion Criteria:

* Patients with systemic bacteremia, positive culture of bacteria of pleural effusion or ascites were excluded from the study because of potential mesh contamination.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-01; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
one-month mortality | one month
  one-month mortality after thoracoscopic mesh repair
three-month mortality | three month
  three-month mortality after thoracoscopic mesh repair

SECONDARY OUTCOMES:
recurrence of hepatic hydrothorax | 20.5 months
  recurrence of hepatic hydrothorax after thoracoscopic mesh repair

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Ming Huang, MD, PhD, Principal Investigator — Department of Surgery, National Taiwan University Hospital

REFERENCES:
- See also: Symptom recovery after thoracic surgery: Measuring patient-reported outcomes with the MD Anderson Symptom Inventory — http://www.ncbi.nlm.nih.gov/pubmed/26088408
- See also: Effect of the amount of intraoperative fluid administration on postoperative pulmonary complications following anatomic lung resections — http://www.ncbi.nlm.nih.gov/pubmed/25304302
- See also: Hepatorenal Disorders — http://www.ncbi.nlm.nih.gov/pubmed/25811649
- See also: Management of refractory hepatic hydrothorax — http://www.ncbi.nlm.nih.gov/pubmed/24811830
- See also: Hepatic hydrothorax — http://www.ncbi.nlm.nih.gov/pubmed/23085762
- See also: Percutaneous transhepatic biliary drainage complicated with hepatic hydrothorax — http://www.ncbi.nlm.nih.gov/pubmed/23312983
- See also: Color Doppler ultrasonography in detecting transdiaphragmatic flow of hepatic hydrothorax: correlation with thoracoscopic findings — http://www.ncbi.nlm.nih.gov/pubmed/19660259
- See also: Thoracoscopic diaphragmatic repair for refractory hepatic hydrothorax: application of pleural flap and mesh onlay reinforcement — http://www.ncbi.nlm.nih.gov/pubmed/16485189
- See also: The morphology of diaphragmatic defects in hepatic hydrothorax: thoracoscopic finding — http://www.ncbi.nlm.nih.gov/pubmed/15999054